CLINICAL TRIAL: NCT04015427
Title: Clinical, Microbiological and Histological Effects of Cemented Implant Restorations. A Cross-over Controlled Clinical Study
Brief Title: Cement Excess at Single Implant Crowns Malmö/Lund
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Folktandvården Skåne AB (Other); Göteborg University (Other); Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-414
Record Dates: First submitted 2018-10-11; First posted 2019-07-11 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Gingivitis and Periodontal Diseases; Tooth Loss
Keywords: cement; dental; implant; implant prosthodontics
MeSH Terms: conditions — Gingivitis; Periodontal Diseases; Tooth Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- screw-retained (Active Comparator): Patients in group A will receive a screw-retained implant crown. Following this first period of 16 weeks, the screw-retained implant crown will be replaced by a new intraorally cemented implant crown. Cement removal will be preformed according to best clinical procedure. These implant crowns will again be left for another period of 16 weeks and followed up for the harvesting of microbiological samples every 8 weeks. After the second 16-week the implant crowns will be removed to evaluate any excess cement. All patients will be fitted with the original screw-retained implant crown. Clinical parameters for inflammation and probing depths will be obtained after each 16 week-period.
  Interventions: Device: implant crown
- cement-retained (Active Comparator): In group B the implant crowns will be incorporated in a reverse pattern. During the first 16 weeks a cemented implant crown will be inserted and any possible cement residues will be removed according to best clinical procedure, while for the second period of 16 weeks patients will be fitted with a screw-retained single implant crown. Again, microbiological and clinical parameters will be obtained at the same intervals as in Group A.
  Interventions: Device: implant crown

INTERVENTIONS:
Device: implant crown — After the second 16 week period the screw-retained crowns will be (re-) inserted in all patients, single tooth x-rays taken and clinical baseline values obtained. Additionally, a soft tissue biopsy will be harvested at the time of insertion of the final screw-retained crown. Patients will be followed up for another 16-week period.

SUMMARY:
Abstract

Aim:

The primary aim of this study is to test whether or not cement residues in the submucosal environment of implants lead to a change in the microbiota and induce inflammation of the periimplant tissues.

Material and Methods:

24 patients in need of a single tooth replacement will be enrolled in this cross-over controlled clinical study. All patients will receive a two-piece dental implant, which will be restored with both a cemented and a screw-retained single crown. At the time of impression taking, patients will be randomized into two groups.

Patients in group A will receive a screw-retained crown. Every 8 weeks microbiological samples using sterile paper points will be collected and analyzed for bacterial content by real-time PCR. Additionally, two host markers (MMP8, IL-1ß) will be determined by ELISA. Following this first period of 16 weeks, the screw-retained crown will be replaced by a new intraorally cemented crown. Cement removal will be preformed according to best clinical procedure. These crowns will again be left for another period of 16 weeks and followed up for the harvesting of microbiological samples every 8 weeks. After the second 16-week the crowns will be removed to evaluate any excess cement. All patients will be fitted with the original screw-retained crown. Clinical parameters for inflammation and probing depths will be obtained after each 16 week-period.

In group B the crowns will be incorporated in a reverse pattern. During the first 16 weeks any possible cement residues will be removed according to best clinical procedure, while for the second period of 16 weeks patients will be fitted with a screw-retained single crown. Again, microbiological and clinical parameters will be obtained at the same intervals as in Group A.

After the second 16 week period the screw-retained crowns will be (re-) inserted in all patients, single tooth x-rays taken and clinical baseline values obtained. Additionally, a soft tissue biopsy will be harvested at the time of insertion of the final screw-retained crown. Patients will be followed up for another 16-week period.

ELIGIBILITY:
Inclusion Criteria:

* - patient older than 18 years
* systemically healthy subject
* periodontally healthy individuals
* absence of peri-implantitis
* no bone loss
* good oral hygiene (PCR ≤ 20%)
* healthy periodontal tissues (BoP≤ 20%)
* patients with a single tooth gap in the posterior area of either jaw (premolars and molars)
* at least 8mm in mandible; at least 6mm in maxilla (summers technique)

Exclusion Criteria:

* - ongoing periodontal disease
* bruxism
* unwilling to comply with study procedures
* heavy smokers (≥10 cig/d)
* ongoing periodontitis/implantitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Analysis of microbiological parameters | Change BL to 16 weeks post-restoration
  Change relative percentage of gram-negative microorganisms

SECONDARY OUTCOMES:
Histomorphometric analysis | 32 weeks after BL
  A soft tissue biopsy will be harvested at the time of insertion of the final screw-retained implant crown in all patients. The biopsies will be used for histomorphometric measurements.
Immunohistologic analysis - putative periodontal pathogens | 32 weeks after BL
  The biopsies will be used for the determination of inflammation and infection markers applying light-microscopy. Gingival crevicular fluid (GCF) will be collected using standardized filter paper strips. A battery of 10 putative periodontal pathogens will be analyzed using real-time PCR.
Immunohistologic analysis - MMP8 | 32 weeks after BL
  The biopsies will be used for the determination of inflammation and infection markers applying light-microscopy. Gingival crevicular fluid (GCF) will be collected using standardized filter paper strips.
Immunohistologic analysis - IL1ß | 32 weeks after BL
  The biopsies will be used for the determination of inflammation and infection markers applying light-microscopy. Gingival crevicular fluid (GCF) will be collected using standardized filter paper strips.
Analysis of inflammation markers on RNA-basis - (IL-4, IL-3, IL-1alfa, IL-1beta) | 32 weeks after BL
  Tissue samples will further be processed with a (ribonucleic acid) RNA solution to allow for RNA extraction. This will then be analyzed via polymerase chain reaction (PCR) to determine expression patterns of markers such as Interleukin (IL-4, IL-3, IL-1alfa, IL-1beta) and tumor necrose factor (TNF-alfa).
Analysis of inflammation markers on RNA-basis - TNF-alfa | 32 weeks after BL
  Tissue samples will further be processed with a (ribonucleic acid) RNA solution to allow for RNA extraction. This will then be analyzed via polymerase chain reaction (PCR) to determine expression patterns of markers such as Interleukin (IL-4, IL-3, IL-1alfa, IL-1beta) and tumor necrose factor (TNF-alfa).
Clinical parameters - Probing Depth | Every 8 weeks until 48 weeks and again at the 1-year follow-up
  In order to assess the inflammatory status of the peri-implant tissue, different parameters will be assessed: 1) plaque index (dichotomous values) 2) keratinized tissue width (continuous) 3) BOP (dichotomous), 4) PD (continuous), 5) recession (continuous)
Clinical parameters - Bleeding-on-Probing | Every 8 weeks until 48 weeks and again at the 1-year follow-up
  In order to assess the inflammatory status of the peri-implant tissue, different parameters will be assessed: 1) plaque index (dichotomous values) 2) keratinized tissue width (continuous) 3) BOP (dichotomous), 4) PD (continuous), 5) recession (continuous)
Clinical parameters - Plaque Index | Every 8 weeks until 48 weeks and again at the 1-year follow-up
  In order to assess the inflammatory status of the peri-implant tissue, different parameters will be assessed: 1) plaque index (dichotomous values) 2) keratinized tissue width (continuous) 3) BOP (dichotomous), 4) PD (continuous), 5) recession (continuous)

OTHER OUTCOMES:
Determination of additional inflammatory markers - MMP8 | 4 times 8 weeks
  The collected microbiological samples will additionally be analyzed for two host markers (MMP8, IL-1ß) that will be determined by ELISA.
Determination of additional inflammatory markers - IL-1ß | 4 times 8 weeks
  The collected microbiological samples will additionally be analyzed for two host markers (MMP8, IL-1ß) that will be determined by ELISA.
Radiological outcomes | 12 weeks pre-BL, BL and 1year post-BL
  A single-tooth x-ray will be obtained at the time of implant placement and again at abutment connection in order to ensure sufficient osseointegration of the implant before entering the prosthetic phase. At the time of insertion of the respective reconstruction in both groups, another periapical radiograph will be obtained to ensure the fit of the reconstruction and to check for eventual cement residue. A final x-ray will be taken at insertion of the final screw-retained implant crown to serve as baseline regarding marginal bone level at the time of final crown insertion.

CONTACTS AND LOCATIONS:
Locations (1):
- Folktandvården Skåne, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
the scans of the sealed randomization envelopes will be sent to the center in Lund, Sweden whenever a patient is included and ready to take the impression.
  A folder structure on switch drive is set up with the Subject numbers (1-24) in order to upload the CRFs, photographs and X rays.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: mid 2020
Access Criteria: login provided by the study monitor (UZH)
URL: http://drive.switch.ch

DOCUMENTS (1):
  • Study Protocol (2018-05-04): https://cdn.clinicaltrials.gov/large-docs/27/NCT04015427/Prot_000.pdf